CLINICAL TRIAL: NCT00619489
Title: Phase 2, Multiple Dose, Open-Label Study to Determine the Long Term Safety of MLN0002 in Patients With Ulcerative Colitis and Crohn's Disease
Brief Title: Long Term Safety of Vedolizumab (MLN0002) in Patients With Ulcerative Colitis and Crohn's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C13004; U1111-1156-8608 (Registry Identifier: WHO)
Record Dates: First submitted 2008-02-11; First posted 2008-02-21 (Estimated); Results first posted 2014-07-18 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-06

CONDITIONS: Ulcerative Colitis; Crohn's Disease
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease | interventions — vedolizumab; LDP-02

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vedolizumab 2 mg/kg (Experimental): Participants received vedolizumab, 2 mg/kg, intravenously (IV), on Days 1, 15 and 43, and thereafter once every 8 weeks for up to 78 weeks.
  Interventions: Drug: vedolizumab
- Vedolizumab 6 mg/kg (Experimental): Participants received vedolizumab, 6 mg/kg, IV, on Days 1, 15 and 43, and thereafter once every 8 weeks for up to 78 weeks.
  Interventions: Drug: vedolizumab

INTERVENTIONS:
Drug: vedolizumab — Vedolizumab for intravenous (IV) infusion
  Other Names: Entyvio; MLN0002; MLN02; LDP-02

SUMMARY:
This was an open-label study to provide an opportunity for participants with Ulcerative Colitis (UC) who previously completed Study C13002 (NCT01177228), and for treatment-naïve participants with UC or Crohn's Disease (CD) to receive treatment with vedolizumab, and to determine the long term safety of vedolizumab in patients afflicted with these diseases.

DETAILED DESCRIPTION:
This was a phase 2, multiple-dose, open-label study of vedolizumab administered intravenously (IV) every 8 weeks. The study population included treatment-naïve ulcerative colitis (UC) or Crohn's Disease (CD) participants, as well as 38 UC participants who had tolerated vedolizumab well during Study C13002 (NCT01177228).

In the original study protocol, all participants were randomized to receive vedolizumab at doses of either 6 mg/kg or 10 mg/kg. With the implementation of Amendment 1, the assigned doses of vedolizumab were decreased to 2.0 mg/kg and 6.0 mg/kg. To implement the dose changes, instead of randomizing all participants across both doses, those who rolled over from Study C13002 were reassigned to receive the 2.0 mg/kg dose and all participants who entered C13004 naïve to treatment were to receive the 6.0 mg/kg dose, starting on the next scheduled dosing day. Also, if participants assigned to the 2 mg/kg dose experienced flare, they were to receive the higher 6 mg/kg dose.

In the results analyses for this study, participants are grouped according to the lowest dose received, i.e., 2.0 mg/kg or 6.0 mg/kg vedolizumab.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed and active ulcerative colitis (UC) or Crohn's Disease (CD)

  * Crohn's Disease Activity Index (CDAI) Score of 220 - 450 for participants with CD
  * Partial Mayo score of 2 - 7 for participants with UC
* Patient should be appropriate candidate for biologic therapy per guidelines
* Up-to-date on cancer screening
* No severe systemic disease
* Patients with evidence of abscess
* Agree to comply with study procedures including contraception

Exclusion Criteria:

* Low lymphocyte counts
* History of imaging abnormalities, multiple sclerosis (MS), brain tumor or other neurological illness
* Active or recent serious infections
* Recent treatment with biologic (i.e., Remicade) or investigational drug
* Impending surgery
* Any participants with vedolizumab human anti-human antibody (HAHA) titers ≥1:125 or with a previous immediate hypersensitivity reaction during or shortly after vedolizumab infusion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2007-12; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

REFERENCES:
- [Derived] Colombel JF, Sands BE, Rutgeerts P, Sandborn W, Danese S, D'Haens G, Panaccione R, Loftus EV Jr, Sankoh S, Fox I, Parikh A, Milch C, Abhyankar B, Feagan BG. The safety of vedolizumab for ulcerative colitis and Crohn's disease. Gut. 2017 May;66(5):839-851. doi: 10.1136/gutjnl-2015-311079. Epub 2016 Feb 18. PMID 26893500

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 14 investigative sites in Canada and Russia, between 07 December 2007 and 31 March 2010.
Pre-assignment Details: Treatment-naïve ulcerative colitis (UC) or Crohn's Disease (CD) participants were assigned to receive 6.0 mg/kg vedolizumab. Participants who rolled over from Study C13002 (NCT01177228) were assigned to receive 2.0 mg/kg vedolizumab.
Period: Overall Study
Arm/Group | Vedolizumab 2 mg/kg | Vedolizumab 6 mg/kg
Started | 37 | 35
Completed | 14 | 1
Not Completed | 23 | 34
Not completed — Adverse Event | 0 | 7
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lack of Efficacy | 0 | 11
Not completed — Rolled over to Study C13008 (NCT00790933 | 22 | 15

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set defined as all enrolled participants who received at least 1 dose of study drug. Patients were analyzed based on the lowest dose they received.
  Baseline is the time closest to, but before, the start of study drug administration; for participants who rolled over from Study C13002 Baseline data are from the C13002 dataset.
Groups:
- Total: Total of all reporting groups
Arm/Group | Vedolizumab 2 mg/kg | Vedolizumab 6 mg/kg | Total
Number analyzed (Participants) | 37 | 35 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.0 (11.06) | 42.1 (15.79) | 42.1 (13.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 22 | 43
  Male | 16 | 13 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 37 | 34 | 71
  Unknown or Not Reported | 0 | 1 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  White | 37 | 34 | 71
  American Indian or Alaskan Native | 0 | 1 | 1
Height [Mean (Standard Deviation); unit: cm] | 168.9 (8.83) | 168.4 (11.49) | 168.7 (10.14)
Weight [Mean (Standard Deviation); unit: kg] | 77.03 (17.620) | 70.81 (17.820) | 74.01 (17.868)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 27.04 (6.045) | 24.86 (5.286) | 25.98 (5.754)
Body Surface Area (BSA) [Mean (Standard Deviation); unit: m^2] | 1.89 (0.233) | 1.81 (0.270) | 1.85 (0.253)
Inflammatory Bowel Disease Type [Number; unit: participants]
  Crohn's Disease | 0 | 19 | 19
  Ulcerative Colitis | 37 | 16 | 53

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An adverse event (AE) is any untoward medical occurrence in a patient administered a pharmaceutical product, which does not necessarily have a causal relationship with the treatment. The investigator systematically collected information adequate to determine both the outcome and severity of the AE, and whether or not it was drug-related or met the criteria for classification as a serious adverse event (SAE). An SAE was defined as an AE that resulted in (or posed risk for) death, inpatient hospitalization (or prolonging hospitalization), or congenital, persistent or significant disability/incapacity.
  The intensity for each AE was defined according to the following criteria:
  Mild: Awareness of sign or symptom, but easily tolerated; Moderate: Discomfort enough to cause interference with normal daily activities; Severe: Inability to perform normal daily activities.
Time Frame: From Day 1 to Day 637
Population: Safety analysis set, defined as all enrolled participants who received at least 1 dose of study drug. Analysis was based on the lowest dose received, rather than dose at randomization.
Measure: Number; unit: participants
Arm/Group | Vedolizumab 2 mg/kg | Vedolizumab 6 mg/kg
Number analyzed (Participants) | 37 | 35
participants
  Any Adverse Event | 21 | 35
  Severe Adverse Event | 2 | 9
  Drug-related Adverse Event | 5 | 21
  Adverse Event Resulting in Discontinuation | 0 | 7
  Serious Adverse Event | 3 | 7
  Drug-related Serious Adverse Event | 1 | 4
  Serious Adverse Event Resulting in Discontinuation | 0 | 5
  On-study Deaths | 0 | 0

2. Primary Outcome: Number of Participants With Clinically Significant Laboratory Findings
Description: Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) are enzymes in the blood.
Time Frame: through Day 637
Population: Safety analysis set
Measure: Number; unit: participants
Arm/Group | Vedolizumab 2 mg/kg | Vedolizumab 6 mg/kg
Number analyzed (Participants) | 37 | 35
participants
  Anemia | 3 | 0
  White Blood Cells Increased | 0 | 1
  White Blood Cells Decreased | 0 | 1
  C-reactive Protein Increased | 1 | 0
  Hypokalemia | 0 | 2
  Hypomagnesemia | 0 | 1
  Hepatic enzyme increased | 0 | 1
  ALT and AST Increased | 0 | 1

3. Primary Outcome: Number of Participants With Signs and Symptoms of Progressive Multifocal Leukoencephalopathy (PML)
Description: At every visit, before receiving study treatment participants were evaluated by clinic staff for signs of PML using a PML symptom checklist.
Time Frame: through Day 637
Population: Safety analysis set
Measure: Number; unit: participants
Arm/Group | Vedolizumab 2 mg/kg | Vedolizumab 6 mg/kg
Number analyzed (Participants) | 37 | 35
participants | 0 | 0

4. Primary Outcome: Number of Participants With Human Anti-human Antibodies (HAHA)
Time Frame: Samples collected prior to dosing on Days 1, 43, 155, 267, 379, 491, and 637.
Population: Safety analysis set
Measure: Number; unit: participants
Arm/Group | Vedolizumab 2 mg/kg | Vedolizumab 6 mg/kg
Number analyzed (Participants) | 37 | 35
participants | 2 | 1

5. Secondary Outcome: Serum Concentration of Vedolizumab Before Dosing
Description: Vedolizumab serum concentrations were measured from serum samples collected for pharmacokinetic (PK) analysis within 2 hours prior to dosing. The original protocol specified that PK parameters, including but not limited to minimum plasma concentration (Cmin), were to be estimated; however, due to intrapatient dose modification with Amendment 1, it was no longer feasible to perform a full PK parameter estimation. The summaries of pre-infusion data (i.e., trough levels) are presented at time points where at least 50% of participants had quantifiable vedolizumab concentrations, using a value of 0 for results below a measurable range. This provides information on the pharmacokinetic behavior of vedolizumab when administered as long-term therapy.
Time Frame: Days 43, 99, 155 and 267, predose
Population: The PK Population included all participants who received at least 1 dose of vedolizumab and had sufficient blood sampling for estimation of PK parameters. Participants without dose modification and with available serum concentration data at each time point (indicated by "n") are included.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Vedolizumab 2 mg/kg | Vedolizumab 6 mg/kg
Number analyzed (Participants) | 27 | 19
μg/mL
  Day 43 (n=27, 19) | 25.2 (6.68) | 76.2 (36.9)
  Day 99 (n=24, 18) | 11.2 (4.33) | 32.5 (20.5)
  Day 155 (n=26, 17) | 8.40 (3.65) | 26.4 (17.7)
  Day 267 (n=26, 12) | 7.40 (3.18) | 25.2 (11.7)

6. Secondary Outcome: Saturation of Receptors by Vedolizumab Before Dosing on Days 1, 43, 99, 155 and 267 by ACT-1 Assay
Description: The target of vedolizumab is α4β7 integrin, a receptor found on inflammatory immune cells that guides these inflammatory cells to the gut and binds to the Mucosal Addressin Cell Adhesion Molecule-1 (MAdCAM-1) on gut endothelial cells. The extent of the α4β7 receptor saturation by vedolizumab was assessed using the ACT-1 binding interference assay. ACT-1 is a mouse antibody similar to vedolizumab that also binds α4β7 integrin. The assay measures the percentage of cells bearing α4β7 that were not saturated with vedolizumab at the time of sampling.
Time Frame: Days 43, 99, 155 and 267, predose
Population: Pharmacodynamic (PD) Population included all participants who received at least 1 dose of vedolizumab and had sufficient blood sampling for estimation of PD parameters. Participants without dose modification and with available PD data at each time point are included.
Measure: Mean (Standard Deviation); unit: % ACT1 binding
Arm/Group | Vedolizumab 2 mg/kg | Vedolizumab 6 mg/kg
Number analyzed (Participants) | 26 | 20
% ACT1 binding
  Day 1 (0, 20) | NA (NA) — Data are not available because only treatment naïve participants were included at the Day 1 time point, and no naïve participants received 2 mg/kg. | 14.6 (4.46)
  Day 43 (26, 19) | 0.277 (0.216) | 0.311 (0.200)
  Day 99 (n=26, 17) | 0.596 (0.690) | 0.288 (0.271)
  Day 155 (n=26, 17) | 0.700 (1.50) | 1.09 (3.31)
  Day 267 (n=25, 12) | 0.276 (0.247) | 0.767 (1.48)

7. Secondary Outcome: Saturation of Receptors by Vedolizumab Before Dosing Using the MAdCAM-1-Fc Assay
Description: The target of vedolizumab is α4β7 integrin, a receptor found on inflammatory immune cells that guides these inflammatory cells to the gut and binds to the mucosal address in cell adhesion molecule-1 (MAdCAM-1) on gut endothelial cells. The extent of the α4β7 receptor saturation by vedolizumab was assessed using the MAdCAM-1-Fc binding interference assay at time points where at least 50% of participants in the analysis set had non-missing results. MAdCAM-1-Fc is a fusion of human MAdCAM-1 with parts of a mouse monoclonal antibody. The assay measures the percentage of cells bearing α4β7 that were not saturated with vedolizumab at the time of sampling.
Time Frame: Days 43, 99, 155 and 267, predose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percent MADCAM binding
Arm/Group | Vedolizumab 2 mg/kg | Vedolizumab 6 mg/kg
Number analyzed (Participants) | 26 | 20
percent MADCAM binding
  Day 1 (n=0, 20) | NA (NA) — Data are not available because only treatment naïve participants were included at the Day 1 time point, and no naïve participants received 2 mg/kg. | 18.5 (5.95)
  Day 43 (n=26, 19) | 0.538 (0.512) | 0.705 (1.29)
  Day 99 (n=26, 16) | 1.22 (1.20) | 0.838 (0.950)
  Day 155 (n=26, 16) | 0.646 (0.673) | 0.369 (0.540)
  Day 267 (n=25, 12) | 1.05 (1.38) | 0.975 (1.55)

ADVERSE EVENTS:
Time Frame: From Day 1 to Day 637
Arm/Group | Vedolizumab 2 mg/kg | Vedolizumab 6 mg/kg
Serious Adverse Events (participants affected / at risk) | 3/37 | 7/35
Other Adverse Events (participants affected / at risk) | 12/37 | 27/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vedolizumab 2 mg/kg (N=37) | Vedolizumab 6 mg/kg (N=35)
Abdominal abscess (Infections and infestations) | 0 | 1
Salmonella sepsis (Infections and infestations) | 0 | 1
Furuncle (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Crohn's disease (Gastrointestinal disorders) | 0 | 1 — Crohn's Disease (CD) relapse among CD patients
Vision blurred (Eye disorders) | 0 | 1
Infusion-related reaction (General disorders) | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Uterine polyp (Reproductive system and breast disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vedolizumab 2 mg/kg (N=37) | Vedolizumab 6 mg/kg (N=35)
Nasopharyngitis (Infections and infestations) | 5 | 7
Influenza (Infections and infestations) | 1 | 3
Upper respiratory tract infection (Infections and infestations) | 1 | 2
Respiratory tract infection viral (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 0 | 2
Viral infection (Infections and infestations) | 0 | 2
Headache (Nervous system disorders) | 2 | 7
Carpal tunnel syndrome (Nervous system disorders) | 2 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 2
Crohn's disease (Gastrointestinal disorders) | 0 | 3 — Crohn's Disease (CD) relapse among CD patients
Nausea (Gastrointestinal disorders) | 0 | 3
Vomiting (Gastrointestinal disorders) | 0 | 3
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 2
Eczema (Skin and subcutaneous tissue disorders) | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2
Influenza like illness (General disorders) | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2
Depression (Psychiatric disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi-site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.